CLINICAL TRIAL: NCT06584448
Title: Role of Acetate in Heavy Drinking
Brief Title: Drinking, Acetate, and Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000035790; R01AA031401 (NIH)
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Alcohol Use, Unspecified; Heavy Drinker; Alcohol Use Disorder, Moderate, in Sustained Remission
Keywords: Brain; Stress; Imaging; Detoxification; Recovery; Sobriety
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcoholic Intoxication; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Light/Non Drinking (LD) (Experimental): Participants will complete an initial telephone screen. Participants found to be potentially eligible will be scheduled for an in-person Intake Session (consisting of an interview, questionnaires, lab work, and a urine drug screen). Participants found to be eligible will be scheduled for an infusion study. Participants will undergo brain imaging with intravenous administration of deuterated sodium acetate. Deuterium is a naturally occurring, non-radioactive substance that allows us to measure rates of metabolism. Neurocognitive tests will be performed to assess the impact of alcohol drinking.
  Interventions: Other: Deuterium Metabolic Imaging with deuterated acetate tracer
- Heavy/Non-Dependent Risky Drinking (HD) (Experimental): Participants will complete an initial telephone screen. Participants found to be potentially eligible will be scheduled for an in-person Intake Session (consisting of an interview, questionnaires, lab work, and a urine drug screen). Participants found to be eligible will be scheduled for an infusion study. Participants will undergo brain imaging with intravenous administration of deuterated sodium acetate. Deuterium is a naturally occurring, non-radioactive substance that allows us to measure rates of metabolism. Neurocognitive tests will be performed to assess the impact of alcohol drinking.
  Interventions: Other: Deuterium Metabolic Imaging with deuterated acetate tracer
- Treatment Seeking (TS) (Experimental): Participants will complete an initial telephone screen. Participants to be potentially eligible will be scheduled for an in-person Intake Session (consisting of an interview, questionnaires, lab work, and a urine drug screen). If found to be eligible participants will be scheduled for an inpatient admission. Participants will take part in an inpatient, medically supervised detoxification. In early sobriety (normally within one week of the last drink) and after approximately one month, participants will undergo brain imaging with intravenous administration of deuterated sodium acetate. Deuterium is a naturally occurring, non-radioactive substance that allows us to measure rates of metabolism. Neurocognitive tests will be performed to assess the impact of alcohol drinking.
  Interventions: Other: Deuterium Metabolic Imaging with deuterated acetate tracer
- Long-Term Recovery (LTS) (Experimental): Participants will complete an initial telephone screen. Participants found to be potentially eligible will be scheduled for an in-person Intake Session (consisting of an interview, questionnaires, lab work, and a urine drug screen). Participants found to be eligible will be scheduled for an infusion study. Participants will undergo brain imaging with intravenous administration of deuterated sodium acetate. Deuterium is a naturally occurring, non-radioactive substance that allows us to measure rates of metabolism. Neurocognitive tests will be performed to assess the impact of alcohol drinking.
  Interventions: Other: Deuterium Metabolic Imaging with deuterated acetate tracer

INTERVENTIONS:
Other: Deuterium Metabolic Imaging with deuterated acetate tracer — Deuterium Metabolic Imaging (DMI) is a method by which Magnetic Resonance Spectroscopy (MRS) is used to map the appearance of deuterium from a tracer source (e.g., deuterated acetate) in products of metabolism. In this case we will map the combination of glutamate and glutamine, called Glx, to serve as a tag to measure the brain's rate of acetate consumption. That is, the more deuterium appears in Glx, the more acetate that part of the brain consumes.
  Other Names: DMI

SUMMARY:
The purpose of this study is to learn how drinking alcohol affects how people experience stress and how that is affected by the body's chemistry. Specifically, the investigators will be studying relationships of drinking and a stress hormone called cortisol. The investigators believe that results will lead us to find more effective ways to help people stop or reduce drinking when participants are drinking at harmful levels.

DETAILED DESCRIPTION:
Brain acetate consumption will be measured with a novel method called Deuterium Metabolic Imaging (DMI), in which sodium acetate that has been labeled with deuterium, a non-radioactive isotope of hydrogen, is administered intravenously over two hours, while Magnetic Resonance Spectroscopy (MRS) is used to map the appearance of the deuterium in glutamate and glutamine regionally through the brain. That combination of glutamate and glutamine, called Glx, serves as a tag to measure the brain's rate of acetate consumption. That is, the more deuterium appears in Glx, the more acetate that part of the brain consumes. In the same people, investigators will perform structural Magnetic Resonance Imaging (MRI) for co-registration with the MRI and assess regional brain volumes. Investigators will also obtain measures of drinking and stress, and will measure participants serum cortisol levels and rates of cortisol turnover. Each set of measures will be compared across groups, and the measurements of acetate uptake will be compared with all other measures for associations.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Medically stable male or female, aged 18-55.
* Able to read, write and complete a multitude of self-assessments in English
* Meets DSM-5 criteria for current Alcohol Use Disorder (AUD)
* Participants who have Alcohol Use Disorder and are actively drinking must be willing to receive (at no cost) inpatient treatment for AUD for a period of up to 30 days. Participants who have been treated for an Alcohol Use Disorder and are now sober three months or longer will NOT be required to go inpatient.

Exclusion Criteria:

* Subjects with any significant current medical conditions (neurological, cardiovascular, endocrine, thyroid, renal, liver), seizures (for LTS subjects only- seizures directly related to alcohol detoxification are not an exclusion) , delirium or hallucinations, or other unstable medical conditions, including HIV.
* Current DSM-5 substance use disorder (other than AUD or tobacco use disorder)
* Any metallic objects implanted in their body which would make imaging unsafe (pacemaker, etc)
* Claustrophobia, or other inability to participate in an MRI
* A positive test result at intake appointment and subsequent appointments on urine drug screens conducted for illicit drugs. (Note: participants will not be paid for study visits if they test positive for an illicit drug and will be immediately excluded from study).
* Women who are pregnant or nursing. Women who have an IUD that would make imaging unsafe.
* Recent taking of medications that may influence study outcomes (e.g., disulfiram, naltrexone, acamprosate, anticonvulsants).
* Subjects likely to exhibit clinically significant alcohol withdrawal during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Conversion of Acetate to Glutamate + Glutamine (Glx) in the Brain | Baseline and for TS, once within approximately one week and again at approximately one month
  DMI data will be acquired during infusions of 2H-labeled Ac, using a 4-Tesla magnet. Deuterium flow from [2,2,2-2H3]Ac to glutamate (Glu) and glutamine (Gln). Ac forms AcetylCoA at a rate CMRAc and is oxidized by astroglia (VtcaA), labeling the small glial Glu pool (5-10% of the total Glu110).Astroglial Glu is converted to Gln and sent to neurons (Vcycle), where it is converted to labeled Glu. It mixes with the large neuronal Glu pool, fed also by unlabeled carbon mostly from glucose via neuronal oxidation (VtcaN), and the diluted Glu is released and taken up by glia for reconversion to Gln. With 2H, the sum of Glu and Gln is detected as [2H]Glx. The faster the rate of acetate consumption, the faster the appearance of [2H]Glx.
Concentration of [2H]Glx in the brain during administration of [2H]acetate | Baseline and for treatment seekers, once after 1 month sober.
  DMI data will be acquired during infusions of 2H-labeled Ac, using a 4-Tesla magnet. Deuterium flow from [2,2,2-2H3]Ac to glutamate (Glu) and glutamine (Gln). Ac forms AcetylCoA at a rate CMRAc and is oxidized by astroglia (VtcaA), labeling the small glial Glu pool (5-10% of the total Glu110).Astroglial Glu is converted to Gln and sent to neurons (Vcycle), where it is converted to labeled Glu. It mixes with the large neuronal Glu pool, fed also by unlabeled carbon mostly from glucose via neuronal oxidation (VtcaN), and the diluted Glu is released and taken up by glia for reconversion to Gln. With 2H, the sum of Glu and Gln is detected as [2H]Glx. The faster the rate of acetate consumption, the faster the appearance of [2H]Glx.

SECONDARY OUTCOMES:
Rate of Cortisol Turnover | Baseline and for treatment seekers, once after 1 month sober.
  Plasma cortisol concentrations and enrichments will be measured in the Chemical Metabolism Core directed by Dr. Kibbey. Crashed plasma samples will be applied to a Phenomenex Kinetex F5 Core-shell LC column (100 x 2.1 mm, 2.6 µm), with 0.3 mL/min linear gradients from 100% aqueous phase (95% water, 5% acetonitrile and 0.1% formic acid) to 100% organic phase (95% acetonitrile, 5% water and 0.1% formic acid) in 20 min. Cortisol ions are measured in both positive and negative MS modes the Sciex TripleTOF 6600 using an information-dependent analysis (IDA) workflow consisting of a TOF MS scan (200 msec) and a high-resolution IDA experiment (70 msec each) monitoring 10 candidate ions per cycle. The ion source conditions are as follows; Ion spray voltage = 5000 V for positive mode and -4500V for negative mode, ion source gas 1 (GS1) = 50, ion source gas 2 (GS2) = 50, curtain gas (CUR) = 30, temperature (TEM) = 400 oC.

OTHER OUTCOMES:
Change in Alcohol and Stress Measures | Baseline and for treatment seekers, once after 1 month sober.
  Measurements of stress and alcohol behaviors, based on questionnaires. Comparison of CMRac with baseline cortisol levels and measures of drinking and craving.Baseline cortisol levels will be compared among groups using a one-way ANOVA followed by post-hoc pairwise tests. Among AD subjects, differences between cortisol levels at 1 week, 1 month, and 3 months will be evaluated with linear mixed models using session (1 week vs. 1 month vs. 3 months). Correlation analysis will be used to examine associations between cortisol levels and levels of CMRac in HPA axis regions, drinking (e.g., # of drinks and drinking days in past 30 days, lifetime consumption), and craving. We will also consider multiple regression models to examine the independent and joint effects of group, cortisol levels, drinking, and craving in predicting CMRac.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Mason, Ph.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - The Anlyan Center, 300 Cedar St., New Haven, Connecticut
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
The data to be shared for all groups are neurocognitive assessments at intake and, for the AUD group, at the one-month time, anatomic MRI, 1H MRS measures, and DMI brain maps of acetate oxidation, and blood cortisol concentrations and isotopic enrichments.
Supporting Information: CSR
Time Frame: The research community will have access to data at publication or at the end of the award, whichever comes first. OpenNeuro standard submission deadlines will be taken into consideration to comply with the timeline requirements. Studies will be uploaded to the OpenNeuro before publication to include their own digital object identifiers (DOI) to aid in findability. We will include that DOI in the relevant publications. OpenNeuro will make decisions about how long to preserve the data. This repository has not deleted any deposited data as far as we know.
Access Criteria: After an optional 36-month embargo period, all datasets are published into the public domain. Prior to being made public, access to a dataset is controlled through strict authentication policies and an isolated storage backend to further guard against unintended access. Metadata describing each dataset snapshot is indexed for searching, and copies of ingested content are provided via persistent Digital Object Identifiers (DOIs) minted for each version of a dataset.